CLINICAL TRIAL: NCT06782282
Title: Real-world Effectiveness of the 20-valent Pneumococcal Conjugate Vaccine (PCV20) Among Medicare Fee-for-service Beneficiaries Aged ≥65 Years in the United States
Brief Title: A Study to Learn About How Well the Prevnar 20 Vaccine Works for Pneumonia in People Who Are 65 Years and Older
Status: Active, not recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B7471043
Record Dates: First submitted 2025-01-03; First posted 2025-01-17 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Community-Acquired Pneumonia (CAP)
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PCV20 Vaccinated: Aged ≥65 years and vaccinated with PCV20 during the study identification period
- PCV20 Unvaccinated: Aged ≥65 years and not vaccinated with PCV20 during the study identification period

SUMMARY:
The purpose of this study is to learn about how well the Prevnar 20 vaccine (PCV20) stops invasive pneumococcal disease (a group of severe infections caused by a bacteria called Streptococcus pneumoniae), pneumococcal pneumonia (a bacterial lung disease caused by the germ Streptococcus pneumoniae), all-cause pneumonia (pneumonia caused by any germ including bacteria, a virus, or a fungus), and lower respiratory tract infection (infection of the lower airways in the lung) in people 65 years and older.

This study will use a database of people who have Medicare insurance with names and other identifying information removed. This study will include people who:

* are 65 years and older,
* live in one of the 50 United States or Washington DC, and
* are enrolled in Medicare Fee-for-Service Parts A and B for at least 1 year.

The study uses data that is already being collected and no treatment or vaccine will be given in the study.

People that fit the description above will be followed in the Medicare database for about two years. Their information will be reviewed to see if they had vaccines for pneumonia or had certain health events, such as pneumonia or lower respiratory tract infection.

The experiences of people that received Prevnar 20 will be compared to the experiences of people that did not receive the vaccine. This will help to show how well Prevnar 20 works at stopping invasive pneumococcal disease, pneumococcal pneumonia, all-cause pneumonia, and lower respiratory tract infection.

DETAILED DESCRIPTION:
Community-acquired pneumonia (CAP) is pneumonia acquired outside of a hospital or within the first 48 hours of hospitalization. It is one of the most common reasons for hospitalization in the US, with up to 10% of patients requiring hospitalization and is the leading cause of infectious disease-related death in the US. Streptococcus pneumoniae remains the leading bacterial cause of CAP, although its incidence has declined over time due to vaccination. Streptococcus pneumoniae is also responsible for Invasive Pneumococcal Disease (IPD).

In 2014, the Advisory Committee in Immunization Practices (ACIP) recommended routine use of the 13-valent pneumococcal conjugate vaccine (PCV13) in series with PPSV23 for all adults aged ≥65 years based on the evidence of PCV13's safety and efficacy against PCV13-type IPD and pneumonia in this age group. A higher valency, 20-valent pneumococcal conjugate vaccine (PCV20) builds on the PCV13 vaccine, and includes seven additional serotypes that cause pneumococcal disease. On October 20, 2021, the ACIP recommended that adults ≥65 years, who had not previously received pneumococcal conjugate vaccine or whose previous vaccination history is unknown may receive PCV20 alone or 15-valent pneumococcal conjugate vaccine (PCV15) in series with PPSV23. On October 19, 2022, the ACIP updated the previous recommendation, recommending that adults who have previously received PCV13 should receive either a dose of the PCV20 or PPSV23.

As a condition of the accelerated approval for PCV20 in June 2021, Pfizer is currently conducting a post-approval confirmatory study to verify and describe the clinical benefit of PCV20 in adults ≥65 years (NCT05452941). In the interim, this study will evaluate the real-world vaccine effectiveness (VE) of PCV20 against IPD, PP, all-cause pneumonia (ACP), and Lower Respiratory Tract Infection (LRTI) among adults aged ≥65 years in Medicare Fee-for-Service (FFS) Parts A, B, and D.

This structured secondary data collection study is a retrospective cohort study using Medicare FFS claims data to estimate real-world PCV20 VE against IPD, PP, ACP, and LRTI among adults aged ≥65 years in the US.

Study analyses will be conducted at the time-segment level, where PCV20 vaccination is a time-varying exposure. In this time-segment design, individuals who receive a PCV20 vaccine during the patient identification period can contribute up to two time segments during the follow-up period: a PCV20 unvaccinated time segment and a PCV20 vaccinated time segment. Each segment will be attributed to the appropriate vaccination exposure status cohort.

Individuals who do not receive a PCV20 vaccine during the patient identification period can contribute a maximum of 1 time segment to the analysis, which will be attributed to the PCV20 unvaccinated cohort. All analyses will be conducted based on time-segment level data.

For PCV20 unvaccinated time segments, individuals will be followed from their unvaccinated index date until the earliest of the following: 1) PCV20 vaccination, 2) PCV13 vaccination, 3) PPSV23 vaccination, 4) PCV15 vaccination, 5) outcome of interest, 6) disenrollment from Medicare FFS Parts A or B, 7) enrollment in Medicare Part C, 8) death, or 9) end of the study period. For PCV20 vaccinated time segments, individuals will be followed from their PCV20 vaccinated index date until the earliest of the following: 1) PCV13 vaccination, 2) PPSV23 vaccination, 3) PCV15 vaccination, 4) second PCV20 vaccination, 5) outcome of interest, 6) disenrollment from Medicare FFS Parts A or B, 7) enrollment in Medicare Part C, 8) death, or 9) end of the study period.

The primary objective is to estimate overall effectiveness of the PCV20 vaccine against three outcome events - first IPD, PP, and ACP due to any serotype - among adults aged ≥ 65 years.

The secondary objective focuses on estimating the overall VE and absolute difference in incidence of PCV20 against LRTI and subgroup VE and absolute difference in incidence stratified by age groups and risk groups. This will involve comparing the time-to-event for LRTI between the vaccinated and unvaccinated using similar methods as described for the primary outcome.

ELIGIBILITY:
Patients from the Medicare database to be included in the analysis must be:

* aged 65 or older as of 28Jan22 (date of 20-valent pneumococcal conjugate vaccine (PCV20)
* residing in one of the 50 US states or Washington DC
* be continuously enrolled in Medicare Fee for Service Parts A and B for 365 days prior to the index date allowing for gaps of up to 45 days (baseline period)

Patients from the Medicare database will be excluded from the analysis if:

* there is a record of death prior to the index date
* the patient was enrolled in Medicare Part C at any point between 28Jan22 and the index date
* the patient received PCV20 before 01Jul22, or the patient received PCV15 prior to the index date

If the patient received the pneumococcal polysaccharide vaccine (PPSV23) within 2 years prior to index date, the corresponding time segment (ie 2 years prior to index date) will be excluded.

If the patient received PCV13 within the past 5 years prior to the index date, the corresponding time segment (ie 5 years prior to index date) will be excluded.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Aged ≥65 years, residing in one of the 50 US states or in Washington, D.C., continuously enrollmed in Medicare FFS Parts A and B for 365 days prior to the index date, allowing for gaps of ≤45 days (baseline period)
Sampling Method: Non-Probability Sample
Enrollment: 22234435 (Actual)
Dates: Start 2025-01-20 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Weighted PCV20 vaccine effectiveness (VE) against Invasive Pneumococcal Disease (IPD) | Time to pneumococcal vaccination, disenrollment from Medicare FFS Parts A or B, enrollment in Medicare Part C, death, or IPD up to 24 months
  Presence of International Classification of Diseases, Tenth Revision, Clinical Modification (ICD-10-CM) codes (1 inpatient or 1 outpatient in any diagnostic position) representing IPD
Weighted PCV20 VE against Pneumococcal Pneumonia (PP) | Time to pneumococcal vaccination, disenrollment from Medicare FFS Parts A or B, enrollment in Medicare Part C, death, or PP up to 24 months
  ICD-10-CM codes (1 inpatient or 1 outpatient in any diagnostic position) representing PP
Absolute difference in the incidence of PP by PCV20 vaccination status | Time to pneumococcal vaccination, disenrollment from Medicare FFS Parts A or B, enrollment in Medicare Part C, death, or PP up to 24 months
  ICD-10-CM codes (1 inpatient or 1 outpatient in any diagnostic position) representing PP
Weighted PCV20 VE against all cause pneumonia (ACP) | Time to pneumococcal vaccination, disenrollment from Medicare FFS Parts A or B, enrollment in Medicare Part C, death, or ACP up to 24 months
  ICD-10-CM codes (1 inpatient or 1 outpatient in any diagnostic position) representing ACP
Absolute difference in incidence of ACP by PCV20 vaccination status | Time to pneumococcal vaccination, disenrollment from Medicare FFS Parts A or B, enrollment in Medicare Part C, death, or ACP up to 24 months
  ICD-10-CM codes (1 inpatient or 1 outpatient in any diagnostic position) representing ACP

SECONDARY OUTCOMES:
Absolute difference in the incidence of IPD by PCV20 vaccination status | Time to pneumococcal vaccination, disenrollment from Medicare FFS Parts A or B, enrollment in Medicare Part C, death, or IPD up to 24 months
  Presence of International Classification of Diseases, Tenth Revision, Clinical Modification (ICD-10-CM) codes (1 inpatient or 1 outpatient in any diagnostic position) representing IPD
Weighted PCV20 VE against Lower Respiratory Tract Infection (LRTI) | Time to pneumococcal vaccination, disenrollment from Medicare FFS Parts A or B, enrollment in Medicare Part C, death, or LRTI up to 24 months
  ICD-10-CM codes (1 inpatient or 1 outpatient in any diagnostic position) representing LRTI
Absolute difference in incidence of LRTI by PCV20 vaccination status | Time to pneumococcal vaccination, disenrollment from Medicare FFS Parts A or B, enrollment in Medicare Part C, death, or LRTI up to 24 months
  ICD-10-CM codes (1 inpatient or 1 outpatient in any diagnostic position) representing LRTI

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer United States, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7471043